CLINICAL TRIAL: NCT02383316
Title: Study of Metabolic Modifications in Children With Noonan Syndrome
Acronym: MetabNoonan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/14/7315; AOL (Other Grant/Funding Number: University Hospital Toulouse, local funding 2014)
Record Dates: First submitted 2014-12-23; First posted 2015-03-09 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2018-02

CONDITIONS: Child Syndrome
Keywords: Insulin sensitivity; Metabolism; Noonan syndrome; Shp2
MeSH Terms: conditions — Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects; Insulin Resistance; Noonan Syndrome | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noonan Syndrome Children (Experimental): Children with Noonan Syndrome will be compared with age- and sex-matched healthy children. We hypothesize than Noonan Syndrome children have an increased insulin sensitivity compared to GHD children.
  Study parameters will be collected including: clinical measurements (height, weight, body mass index, waist circumference, and blood pressure), glucose and insulin levels at baseline and after an oral glucose tolerance test (OGTT), body composition measured by dual-energy x-ray absorptiometry (DXA).
  Interventions: Other: Oral Glucose tolerance test

INTERVENTIONS:
Other: Oral Glucose tolerance test — Oral glucose tolerance test (OGTT): glucose and insulin levels will be measured at time points 0, 90 and 120 min or 30, 60, 90 and 120 after 1.75 g/Kg (max 75 g) glucose administration depending of the patient weight.

SUMMARY:
Noonan syndrome (NS) is a rare genetic disease (incidence 1/2500 live births) characterized by the association of craniofacial manifestations, cardiopathies, short stature, and tumor predisposition. The genetic causes of Noonan Syndrome are mutations of genes involved in the Ras/Mitogen-Activated Protein Kinases (MAPK) pathway, mainly the gene encoding the tyrosine phosphatase Shp2 (50% of patients).Shp2 appears to be involved in many facets of energy metabolism control (glucose homeostasis, adipose tissue function…), through mechanisms that are poorly understood. Several metabolic anomalies (reduced adiposity, improved glucose tolerance) have been recently identified in an original mouse model carrying Shp2 mutation. Moreover, recent clinical survey has shown that adult Noonan Syndrome patients are protected from developping overweight and obesity when compared to the general population. However, the metabolic status associated with Noonan Syndrome condition has not been explored to date.

DETAILED DESCRIPTION:
Differential hormone sensitivity is associated with Noonan Syndrome and participates in the development of some symptoms. The investigators have demonstrated that MAPK upregulation in Noonan Syndrome is responsible for partial growth hormone (GH) insensitivity, and subsequent growth retardation.

Clinical traits evocative of energy metabolism dysfunctions have been recently reported in Noonan Syndrome patients, although the origins and consequences of these metabolic changes have not been documented to date. The aim of this study is to explore the metabolic status of children with Noonan Syndrome.

Children with Noonan Syndrome will be compared with age- and sex-matched healthy children. The investigators hypothesize than Noonan Syndrome children have an increased insulin sensitivity compared to GHD children.

Study parameters will be collected including: clinical measurements (height, weight, body mass index, waist circumference, and blood pressure), glucose and insulin levels at baseline and after an oral glucose tolerance test (OGTT), body composition measured by dual-energy x-ray absorptiometry (DXA).

The study will include only one visit.

ELIGIBILITY:
Inclusion Criteria:

* Noonan syndrome genetically confirmed
* Informed consent obtained from children and parents

Exclusion Criteria:

* Chronic disease associated with variation of insulin sensitivity: body mass
* Treatment associated with variation of insulin sensitivity: corticoid treatment > 5 days preceding the study inclusion
* Tumoral disease (leukemia) in treatment

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity determined from the calculation of the Quantitative insulin sensitivity check index (QUICKI). | T0 on an empty stomach
  Measured at the patient's arrival (TO) from the blood levels of glucose and fasting insulin

SECONDARY OUTCOMES:
Insulin sensitivity determined with HOMA index | T30, T60, T90 and T120 minutes after oral glucose tolerance test
  Glucose and insulin levels will be measured at time points 0, 90 and 120 min (children weigh 17-25kg) or 30, 60, 90 and 120 min (children weigh >25kg) after 1.75g/kg glucose administration (oral glucose tolerance test)
Blood pressure | T0
  These tests will be done on arrival in hospital before the oral glucose tolerance test. Blood pressure is measured after 10 minutes of rest in the elongated child.
Blood level of hemoglobin A1c and ghrelin | T0 on an empty stomach
  Blood sample realised at T0 before the oral glucose tolerance test.
Body composition as fat mass and muscle mass measured by dual-energy x-ray absorptiometry (DXA) | T0
  This test will be realised during hospitalisation day, except if it has been done up to 6 months prior to enrollment.
Body mass index | T0
  This test will be realised during hospitalisation day, at patient arrival.
Waist circumference | T0
  This test will be realised during hospitalisation day, at patient arrival.
Blood level of leptin | T0 on an empty stomach
  Blood sample realised at T0 before the oral glucose tolerance test.
Blood level of ghrelin | T0 on an empty stomach
  Blood sample realised at T0 before the oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Edouard, MD, Principal Investigator — CHU Toulouse, Hôpital des Enfants
Locations (1):
- CHU Toulouse - Hôpital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paccoud R, Saint-Laurent C, Piccolo E, Tajan M, Dortignac A, Pereira O, Le Gonidec S, Baba I, Gelineau A, Askia H, Branchereau M, Charpentier J, Personnaz J, Branka S, Auriau J, Deleruyelle S, Canouil M, Beton N, Salles JP, Tauber M, Weill J, Froguel P, Neel BG, Araki T, Heymes C, Burcelin R, Castan I, Valet P, Dray C, Gautier EL, Edouard T, Pradere JP, Yart A. SHP2 drives inflammation-triggered insulin resistance by reshaping tissue macrophage populations. Sci Transl Med. 2021 Apr 28;13(591):eabe2587. doi: 10.1126/scitranslmed.abe2587. Epub 2021 Apr 28. PMID 33910978